CLINICAL TRIAL: NCT00561002
Title: Annual Study for Serum Collection and Evaluation of Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Influenza Virus Vaccine (2007-2008 Formulation)
Brief Title: Phase IV Trial to Collect Safety Data and Sera for Immunogenicity Testing in Healthy Children Given Fluzone® Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC38
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2009-08-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza Vaccine; Influenza Virus; Orthomyxoviridae Infections; Fluzone®
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine Naive/Inadequately Primed (Experimental): Participants had no more than one previous lifetime dose of influenza vaccine and received two doses of Fluzone®, on Days 0 and 14.
  Interventions: Biological: 2007-2008 Influenza Virus Vaccine
- Influenza Vaccine Primed (Experimental): Participants had previously received 2 injections of Influenza vaccine in the same season and received a single dose of Fluzone® on Day 0.
  Interventions: Biological: 2007-2008 Influenza Virus Vaccine

INTERVENTIONS:
Biological: 2007-2008 Influenza Virus Vaccine — 0.25 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Influenza vaccine Naive/Inadequately Primed
Biological: 2007-2008 Influenza Virus Vaccine — 0.25 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Influenza Vaccine Primed

SUMMARY:
To provide Centers for Biologic Evaluation and Research (CBER) with sera collected from healthy children receiving the 2007-2008 formulation of the inactivated, split-virion influenza vaccine Fluzone® for further study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged ≥ 6 months (24 weeks) to < 36 months (3rd birthday).
* Participant is considered to be in good health on the basis of reported medical history and limited physical examination.
* Participant is available for the duration of the study.
* Parent/legal acceptable representative is willing and able to provide informed consent.
* Parent/legal acceptable representative is willing and able to meet protocol requirements.
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* Reported allergy to egg proteins, chicken proteins, or any other constituent of the vaccine.
* An acute illness with or without fever (For infants/toddlers: temperature ≥ 100.4°F rectal; For children: temperature ≥ 99.5°F oral/axillary) in the 72 hours preceding enrollment in the trial (Enrollment may be deferred).
* Clinically significant findings in vital signs or review of systems (Investigator judgment; defer or exclude).
* Participation in any other interventional clinical trial within 30 days prior to enrollment or planned participation in the study.
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known human immunodeficiency virus (HIV)-positive mother.
* Prior personal history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the Investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Received any vaccinations within the preceding 14 days (enrollment may be deferred).

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 29 October 2007 through 27 November 2007 at 1 US site.
Pre-assignment Details: A total of 34 participants who met the inclusion and exclusion criteria were enrolled, 2 were not vaccinated and excluded from the analysis.
Period: Overall Study
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed
Started | 23 | 9
Completed | 23 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed | Total
Number analyzed (Participants) | 23 | 9 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 9 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 19.8 (8.76) | 24.5 (5.10) | 21.2 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Solicited Injection Site and Systemic Reactions After Vaccination With Fluzone 2007-2008 Formulation
Description: Solicited injection site reactions: Erythema, swelling, pain/tenderness; Solicited systemic reactions: (for infants/toddlers) - fever, irritability, abnormal crying, drowsiness, lost appetite, vomiting; (for children) - fever, headache, malaise, myalgia) Note: Influenza-primed group received only dose 1.
Time Frame: Days 0-3 post-dose
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed
Number analyzed (Participants) | 23 | 9
Participants
  Any Solicited Injection Site Reaction Post-dose 1 | 13 | 4
  Any Tenderness | 9 | 2
  Grd 3 Tenderness (Cries when limb is moved) | 0 | 0
  Any Pain | 3 | 2
  Grd 3 Pain (Incapacitating) | 0 | 0
  Any Redness (> 0.5 cm) | 3 | 0
  Grade 3 Redness (≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 2 | 0
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Injection Site Reaction Post-dose 2 | 7 | 0
  Any Tenderness | 6 | 0
  Grd 3 Tenderness (Cries when limb is moved) | 1 | 0
  Any Pain | 1 | 0
  Grd 3 Pain (Incapacitating) | 0 | 0
  Any Redness (> 0.5 cm) | 0 | 0
  Grade 3 Redness) (≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 0 | 0
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Injection Reaction - Any dose | 14 | 4
  Any Tenderness | 10 | 2
  Grade 3 Tenderness (Cries when limb moved) | 1 | 0
  Any Pain | 3 | 2
  Grade 3 Pain (Incapacitating) | 0 | 0
  Any Redness (> 0.5 cm) | 3 | 0
  Grade 3 Redness (≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 2 | 0
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Systemic Reaction Post-dose 1 | 14 | 6
  Any Fever | 4 | 2
  Grade 3 Fever (>103.1 ºF) | 1 | 0
  Any Vomiting | 1 | 0
  Grade 3 Vomiting (≥ episodes per 24 hr) | 0 | 0
  Any Abnormal Crying | 9 | 2
  Grade 3 Abnormal Crying (> 3 hr) | 0 | 0
  Any Drowsiness | 7 | 3
  Grade 3 Drowsiness (Sleeps most of the time) | 0 | 0
  Any Loss of Appetite | 7 | 1
  Grade 3 Loss of Appetite (Refuses most feeds) | 0 | 0
  Any Irritability | 11 | 3
  Grade 3 Irritability (Inconsolable) | 1 | 0
  Any Headache | 0 | 0
  Grade 3 Headache (Prevents daily activities) | 0 | 0
  Any Myalgia | 2 | 0
  Grade 3 Myalgia (Prevents daily activities) | 0 | 0
  Any Malaise | 3 | 3
  Grade 3 Malaise (Prevents daily activities) | 0 | 0
  Any Solicited Systemic Reaction Post-dose 2 | 11 | 0
  Any Fever | 3 | 0
  Grade 3 Fever (> 103ºF) | 0 | 0
  Any Vomiting | 0 | 0
  Grade 3 Vomiting (≥ 6 episodes per 24 hr) | 0 | 0
  Any Abnormal Crying | 5 | 0
  Grade 3 Abnormal Crying (>3 hr) | 0 | 0
  Any Drowsiness | 5 | 0
  Grade 3 Drowsiness (Sleeps most of time) | 0 | 0
  Any Loss of Appetite | 3 | 0
  Grade 3 Loss of Appetite (Refuses most feeds) | 0 | 0
  Any Irritability | 7 | 0
  Grade 3 Irritability (Inconsolable) | 0 | 0
  Any Headache | 0 | 0
  Grade 3 Headache (Prevents daily activities) | 0 | 0
  Any Myalgia | 1 | 0
  Grade 3 Myalgia (Prevents daily activities) | 0 | 0
  Any Malaise | 1 | 0
  Grade 3 Malaise (Prevents daily activities) | 0 | 0
  Any Solicited Systemic Reaction (Any dose) | 16 | 6
  Any Fever | 6 | 2
  Grade 3 Fever (> 103.1 ºF) | 1 | 0
  Any Vomiting | 1 | 0
  Grade 3 Vomiting (≥ 6 episodes per 24 hr) | 0 | 0
  Any Abnormal Crying | 10 | 2
  Grade 3 Abnormal Crying (> 3 hr) | 0 | 0
  Any Drowsiness | 8 | 3
  Grade 3 Drowsiness (Sleeps most of the time) | 0 | 0
  Any Loss of Appetite | 9 | 1
  Grade 3 Loss of Appetite (Refuses most feeds) | 0 | 0
  Any Irritability | 12 | 3
  Grade 3 Irritability (Inconsolable) | 1 | 0
  Any Headache | 0 | 0
  Grade 3 Headache (Prevents activities) | 0 | 0
  Any Myalgia | 2 | 0
  Grade 3 Myalgia (Prevents activities) | 0 | 0
  Any Malaise | 3 | 3
  Grade 3 Malaise (Prevents activities) | 0 | 0

2. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Hemagglutinin Antibodies Pre- and Post-Fluzone® Vaccination
Time Frame: Day 0 and Day 14 after last dose of Fluzone
Population: The Geometric Mean Titers analysis were on the per-protocol immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed
Number analyzed (Participants) | 16 | 6
Titers
  A/Solomon Islands/3/2006 IVR-145 (H1N1) Pre-dose | 8.31 [4.48 to 15.4] | 5.61 [4.17 to 7.55]
  A/Solomon Islands/3/2006 IVR-145 (H1N1) Post-dose | 397 [243 to 649] | 180 [63.1 to 511]
  A/Wisconsin/67/2005 (X-161B) (H3N2) Pre-dose | 10.7 [5.11 to 22.5] | 59.9 [8.94 to 402]
  Wisconsin/67/2005 (X161B) (H3N2) Post-dose | 260 [168 to 401] | 479 [200 to 1148]
  B/Malaysia Split/2506/2004 Pre-dose | 12.3 [5.96 to 25.4] | 13.3 [3.92 to 45.5]
  B/Malaysia Split/2506/2004 Post-dose | 186 [72.6 to 477] | 180 [70.2 to 459]

3. Other Pre Specified Outcome: Percentage of Participants With at Least a 40 Serum Hemagglutination Inhibition Antibody Titers Post-Vaccination (Seroprotection)
Description: Seroprotection was defined as a serum hemagglutination inhibition antibody titer ≥40.
Time Frame: Day 14 post-vaccination
Population: The serum hemagglutination inhibition antibody analysis were on the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed
Number analyzed (Participants) | 16 | 6
Percentage of Participants
  A/Solomon Islands/3/2006 IVR-145 (H1N1) | 100 | 83
  A/Wisconsin/67/2005 (X-161B) (H3N2) | 100 | 100
  B/Malaysia Split/2506/2004 | 81 | 100

4. Other Pre Specified Outcome: Seroconversion Rates for Each Influenza Antigen Post-Vaccination
Description: Seroconversion was defined as a post-vaccination titer ≥ 40 for participants with a titer < 10 on Day 0 and a ≥4-fold increase for participants with a titer ≥ 10 on Day 0.
Time Frame: Day 14 post-vaccination
Population: The seroconversion analysis were on the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed
Number analyzed (Participants) | 16 | 6
Percentage of Participants
  A/Solomon Islands/3/2006 IVR-145 (H1N1) | 100 | 83
  A/Wisconsin/67/2005 (X-161B) (H3N2) | 79 | 67
  B/Malaysia Split/2506/2004 | 80 | 100

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 14 days post-vaccination (Influenza Vaccine Primed group) or 42 days post-vaccination (Influenza Vaccine Naïve/Inadequately Primed group)
Arm/Group | Influenza Vaccine Naive/Inadequately Primed | Influenza Vaccine Primed
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/9
Other Adverse Events (participants affected / at risk) | 12/23 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine Naive/Inadequately Primed (N=23) | Influenza Vaccine Primed (N=9)
Injection site tenderness (General disorders) | 10 | 2
Injection site pain (General disorders) | 3 | 2
Injection site redness (General disorders) | 3 | 0
Injection site swelling (General disorders) | 2 | 0
Pyrexia (General disorders) | 6 | 2
Crying (Psychiatric disorders) | 10 | 2
Somnolence (Nervous system disorders) | 8 | 3
Anorexia (Metabolism and nutrition disorders) | 9 | 1
Irritability (Psychiatric disorders) | 12 | 3
Malaise (General disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications